CLINICAL TRIAL: NCT06368076
Title: High-intensity Interval Training in Patients With Spinal Muscular Atrophy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, John Vissing, Prof. MD., Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-23065096
Record Dates: First submitted 2024-02-29; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Spinal Muscular Atrophy
Keywords: Wheelchair cycle exercise
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — High intensity interval training on a bike or pedaltrainer from the wheelchair.

SUMMARY:
Patients with spinal muscular atrophy who are wheelchair users often experience lower back - and gluteal pain, reduced sleep quality, constipation and reduced quality of life - symptoms that regular exercise could potentially alleviate. However, only very little research has been done on exercise for patients who are wheelchair users. The aim of this study is to explore the impact of cycle exercise on patients with spinal muscular atrophy.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a neuromuscular disease affecting the motor neurons of the spinal cord that innervate the skeletal muscles, leading to progressive muscle atrophy and weakness. Consequently, many patients end up having to use a wheelchair from an early age.

Besides the impaired motor function, patients with SMA can also experience a variety of symptoms associated with their disease, a sedentary lifestyle and physical inactivity such as lower back and leg pain, obstipation, reduced sleep quality and impacted quality of life.

Training can help alleviate these symptoms in patients with neuromuscular diseases. However, there isn´t any validated way for patients with SMA to train as of today.

Research has shown that high-intensity interval training (HIIT) has been well tolerated among patients with SBMA, a disease resembling SMA with patients tolerating this form for training well.

The aim of this study is to investigate:(1) if HIIT could be exercise modality in SMA patients (2) and to see what positive effects exercise has for their impaired motor function and related challenges.

The investigators will test the participants at baseline, which will be followed by a 8-week control period. After the control period the participants will be tested again before the intervention period.

During the intervention period the participants will have to train 5 times a week for 10 minutes. After the intervention period, there will be a final test day, where the final results will be compared with those from the baseline.

ELIGIBILITY:
Inclusion Criteria:

* Spinal muscular atrophy
* Age: over 15 years

Exclusion Criteria:

* Competing disorders (as arthritis) or other muscle disorders as well as heart- or lung related issues.
* Current psychiatric treatment
* Unable to use the cycle ergometer due to contractures

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaire on fatigue | 5 minutes
  The Multidimensional Fatigue Inventory (MFI-20) will be used. It measures fatigue in 5 different domains comprised of 4 items each with values ranging from 1 to 5. A higher score indicates more fatigue. Each domain is scored individually, ranging from 4 points (best outcome) to 20 points (worst outcome).
Questionnaire on pain. | 5 minutes
  A visual pain score for leg and lower back pain with 3 questions with scores ranging from 1 to 10 each, 10 being the worst pain imaginable, will be used.
Questionnaire on constipation | 5 minutes
  A questionnaire made from the Danish definition of constipation will be used. Four questions will be answered "yes" or "no".
Questionnaire on quality of life | 10 minutes
  A QoL that has been used in former studies will be used. 16 questions with scores ranging from 1 (very unsatisfied) to 7 (very satisfied) will be scored.
Questionnaire on sleep quality | 10 minutes
  Minimum Score = 0 (better); Maximum Score = 21 (worse) Interpretation: TOTAL < 5 associated with good sleep quality TOTAL > 5 associated with poor sleep quality Minimum Score = 0 (better); Maximum Score = 21 (worse) Interpretation: TOTAL < 5 associated with good sleep quality TOTAL > 5 associated with poor sleep quality Minimum score is 0, maximum score is 21. Total over 5 is associated with good sleep quality and under 5 associated with poor sleep quality.

SECONDARY OUTCOMES:
Blood sample | 2 minutes
  Change in blood sample for blood lipids, mmol/l
Blood sample | 2 minutes
  Change in blood sample for HbA1C, mmol/mol
Blood sample | 2 minutes
  Change in blood sample for Creatine kinase, U/I. This will be monitored before, in the middle and after the exercise period as a safety measure.
Blood sample | 2 minutes
  Change in blood sample for fasting blood glucose, in mmol/L
Blood sample | 2 minutes
  Change in blood sample for fasting insulin, in pmol/L.
Blood sample | 2 minutes
  Change in blood sample for fasting c-peptide, in pmol/L.
Blood sample | 2 minutes
  Change in blood sample for ALT (liver parameter) in U/L
Blood sample | 2 minutes
  Change in blood sample for AST (liver parameter) in U/L
Blood sample | 2 minutes
  Change in blood sample for alkaline phosphatase (liver parameter) in U/L
Blood sample | 2 minutes
  Change in blood sample for bilirubin (liver parameter) in umol/L
MRI scan liver size | 5 minutes
  Assessment of liver size
MR-elastography | 5 minutes
  Assessment of liver fibrosis (assessed by MR-elastography)
MRI scan liver steatosis | 5 minutes
  Assessment of liver steatosis
Ultrasound scan | 15 minutes
  Additional assessment of liver size, fibrosis and steatosis
MRI scan | 15 minutes
  Assessment of full body muscle size
MRI scan | 15 minutes
  Assessment of muscle degeneration and subsequent fat replacement (using Dixon method to visualise fat in an optimal way)
Exercise test | 7 minutes
  Change in time to cycle X km in minutes
Motorscore | 20 minutes
  Change in motor function score, using the Motor Function Measurement (MFM-32). Assesses motor function in 3 domains, 32 two items in total. A higher score in each domain indicates better function.

CONTACTS AND LOCATIONS:
Overall Officials: John Vissing, prof. MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided